CLINICAL TRIAL: NCT04648306
Title: Restore EF Observational Study (in High-risk PCI)
Brief Title: Restore EF Observational Study
Status: Completed | Type: Observational
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: V1-07012019
Record Dates: First submitted 2020-11-17; First posted 2020-12-01 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Disease; Unstable Angina; Angina, Stable; NSTEMI - Non-ST Segment Elevation MI
Keywords: Impella; Hemodynamic Mechanical Support; Left ventricular ejection fraction; Surgical turndown; High Risk PCI
MeSH Terms: conditions — Coronary Artery Disease; Angina, Unstable; Angina, Stable; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Impella cohort: Single arm study of patients who underwent non-emergent percutaneous coronary intervention with prophylactic Impella support
  Interventions: Device: Prophylactic Impella support for a non-emergent PCI

INTERVENTIONS:
Device: Prophylactic Impella support for a non-emergent PCI — Impella percutaneous mechanical circulatory support is placed via the femoral or axillary artery prior to a non-emergent PCI in patients at high risk for periprocedural complications including hemodynamic collapse.

SUMMARY:
A multi-center, prospective, observational, non-interventional single arm, study of the intermediate-term clinical outcomes collected from electronic health records of high-risk patients which have previously undergone standard of care prophylactic Impella support for a non-emergent percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
1. Hypothesis The prophylactic use of Impella 2.5 or CP heart pumps during a non-emergent PCI in hemodynamically stable patients at high-risk for periprocedural complications during the procedure is associated with a significant improvement in the patient's LVEF and clinical status (heart failure symptoms and hospital readmissions) in the intermediate-term follow-up period post-ProPCI
2. Objectives The primary objective of this study is to assess the patient's LVEF at 90 days post-ProPCI (60 to 180 days window) as assessed in routine clinical practice and collected from EHR by clinical investigators.

   The secondary objective of the study is to assess the potential association between the completeness of revascularization and the clinical status at 90 days post-ProPCI (60-180 days window). Clinical status includes NYHA heart failure functional class and hospital readmission.
3. Sample Size: The study will enroll more than 1,000 patients at up to 30 investigational sites with experienced Impella operators (≥ 25 cases).
4. Primary Endpoint: Subject's LVEF at 90 days post-ProPCI (60 to 180 days window) collected from the subject's EHR.
5. Secondary Endpoints:

   * Completeness and extent of revascularization
   * NYHA functional class at 90 days post-ProPCI (60 to 180 days window)
   * Readmission at 90 days post-ProPCI (60 to 180 days window)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Subject has previously undergone (≥ 60 days) an Impella Protected PCI (ProPCI) at a study site as identified in the Impella quality (IQ) assurance database (patients who expired or were lost to follow-up prior to opening of the follow-up study window (day 60 post Impella protected PCI) will not be included in the study

Exclusion Criteria:

* Subject with cardiogenic shock at the time of Impella insertion. Cardiogenic shock defined as: systemic hypotension (systolic blood pressure (SBP) <90 mmHg or the need for inotropes/pressors to maintain a SBP >90mmHg)
* Subject with ST elevation myocardial infarction at the time of Impella insertion.
* Subject underwent coronary bypass surgery after the index Impella ProPCI
* Subject underwent repeat revascularization with PCI after the index Impella ProPCI
* Subject underwent other cardiac procedures including valve therapies (surgical or percutaneous) after the index Impella ProPCI
* Subject underwent cardiac resynchronization therapy (CRT) initiated after the index Impella ProPCI
* Any known medical condition with a life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet all the inclusion criteria and none of the exclusion criteria will be enrolled in the study.
  Patients in whom prophylactic hemodynamic support with Impella was used during a non-emergent PCI will be evaluated for study participation at 60 days post index PCI procedure with Impella. In this study the index procedure is designated as Impella Protected PCI (ProPCI). Patients with cardiogenic shock and/or ST elevation myocardial infarction (STEMI) at the time of Impella initiation will not be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 90 days post Protective PCI (60 to 180 days window)
  Left ventricular ejection fraction (LVEF) %

SECONDARY OUTCOMES:
Survival Rate | 90 days post Protected PCI (60 to 180 days window)
  Survival rate post non-emergent percutaneous coronary intervention (ProPCI)
NYHA Functional Class | 90 days post Protected PCI (60 to 180 days window)
  New York Heart Association (NYHA) functional class
Readmission | 90 days post Protected PCI (60 to 180 days window)
  Readmission post non-emergent percutaneous coronary intervention (ProPCI)

CONTACTS AND LOCATIONS:
Overall Officials: Thom Dahle, MD, Study Chair — Saint Cloud Hospital; Jason Wollmuth, MD, Study Chair — Providence Health & Services; Lynn Morris, MD, Study Chair — East Carolina University; Craig Thompson, MD, Study Chair — NYU Langone
Locations (21):
- United States (21):
  - St. Joseph's Medical Center, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - Arkansas Cardiology P.A., North Little Rock, Arkansas
  - Northwest Medical Center, Springdale, Arkansas
  - Loma Linda University Medical, Loma Linda, California
  - UCSD Medical Center, San Diego, California
  - Advent Health, Daytona Beach, Florida
  - NorthShore University HealthSystem, Skokie, Illinois
  - Genesis Medical Center, Davenport, Iowa
  - Baptist Healthcare System, Lexington, Kentucky
  - Lafayette General Medical Center, Houma, Louisiana
  - Mercy Hospital, Coon Rapids, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - NYU Langone Medical Center, New York, New York
  - Vidant Medical Center, Greenville, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Presbyterian Hospital Dallas, Arlington, Texas
  - Kingwood Medical Center, Kingwood, Texas
  - Sentara Healthcare, Norfolk, Virginia